CLINICAL TRIAL: NCT02300155
Title: Improving Multivitamin Supplementation to Pregnant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Duchesnay Inc. (Industry)
Responsible Party: Principal Investigator, Gideon Koren, Director of MotherRisk Program, Clinical Pharmacology and Toxicology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000005135
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy; Morning Sickness; Nausea; Vomiting; Hyperemesis Gravidarum
Keywords: Pregnancy; Morning Sickness; nausea and vomiting; hyperemesis gravidarum; perinatal vitamins
MeSH Terms: conditions — Morning Sickness; Nausea; Vomiting; Hyperemesis Gravidarum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PregVit® (Experimental): Women will be randomized to the '35 mg' group, who will start supplementation with PregVit® (low iron content, small size)
  Interventions: Drug: Pregvit®
- Orifer F® (Active Comparator): Women will be randomized to the '60 mg' group, who will start supplementation with Orifer F® (high iron content, small size).
  Interventions: Drug: Orifer F®

INTERVENTIONS:
Drug: Pregvit® — Women were randomized to one of two groups. An information package was mailed to each woman, instructing her to commence supplementation with her assigned prenatal multivitamin, according to the product's standard dosing -twice daily for '35 mg' group
  Other Names: Dietary supplement-prenatal multivitamin
  Arms: PregVit®
Drug: Orifer F® — Women were randomized to one of two groups. An information package was mailed to each woman, instructing her to commence supplementation with her assigned prenatal multivitamin, according to the product's standard dosing-once daily for '60 mg' group
  Other Names: Dietary supplement-prenatal multivitamin
  Arms: Orifer F®

SUMMARY:
The purpose of this study is to compare the tolerability of Pregvit® to a common prenatal vitamin (Orifer® F) among pregnant women with morning sickness or those suffering from a variety of conditions.

DETAILED DESCRIPTION:
Presently, there is a large choice of perinatal vitamins on the market. Materna® is taken by 70% of Canadian women. A recent study by the investigators team has shown that up to 35%-53% of women with moderate to severe morning sickness discontinue their Materna®. One main reason is that its large size causes difficulties in swallowing, which prompts women to stop taking the drug. The second main reason for stopping is gastrointestinal adverse effects from the iron content, which causes nausea, vomiting and constipation.

A new periconceptional multivitamin supplement, Pregvit®, was introduced to the market in September 2003 by the Canadian company Duchesnay Inc. with the aim of trying to overcome the disadvantages of the existing multivitamin supplements. PregVit® is a prenatal multivitamin that contains 35 mg elemental iron, as ferrous fumarate. It is formulated into 2 small tablets (each tablet:16 mm × 9 mm × 4 mm), containing different vitamins and minerals, particularly separating the iron (morning tablet) from the calcium (evening tablet) to optimize iron absorption. The use of PregVit® requires a physician's prescription.

Since Materna® or other generic products are the most commonly used non-prescription (i.e. over-the-counter) prenatal multivitamins, they were not selected for comparison in the study because enrolled subjects who had discontinued a prenatal multivitamin most likely had discontinued any one of them. Ethically, subjects in this situation cannot be randomized to resume Materna® or another generic prenatal multivitamin.

Instead, Orifer F® was selected as the small-tablet prenatal multivitamin (one tablet: 5 mm radius, 5 mm thickness), containing a high iron content (60 mg elemental iron as ferrous sulphate). It is taken daily as a single tablet and the use of Orifer F® does not require a physician prescription (i.e. over-the-counter).

Comparing tolerability of PregVit® to Orifer F® would address separation of the potential effect of iron content from that of tablet size on multivitamin tolerability among pregnant women and women suffering from morning sickness or those suffering from a variety of conditions such as, Crohn's Disease, Ulcerative Colitis, Peptic-Duodenal Ulcer, Irritable Bowel Syndrome, Celiac Disease, as well as anemia or hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

Any woman who discontinued her standard vitamins due to gastrointestinal symptoms or due to the tablet size, with one ofthe following conditions:

* Morning sickness.
* Gastrointestinal disorders: Crohn's disease, ulcerative colitis, peptic or duodenal ulcer, irritable colon, celiac disease.
* Iron deficiency anemia.
* Hypothyroidism.
* Depression.

Exclusion Criteria:

* Women who do not agree to consent to this protocol.
* Women with a known hypersensitivity to any of the ingredients of Pregvit®, or Orifer® F.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1370 (Actual)
Dates: Start 2004-10; Primary Completion 2006-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The difference in rates of ability to take multivitamin [either Pregvit® or Orifer®F] | Study completion was defined as completing monthly telephone interviews (when possible) to document pill intake and adverse events up until the end of pregnancy (i.e. 36 weeks gestation or further).
  Rates of adherence and adverse events will be compared by using chi-squared tests, as appropriate. Adherence will be also compared between the 2 treatment groups through Kaplan-Meier survival curves in 2 ways. The first survival curve analysis will compare the proportion of women with standard adherence (i.e. at least 80% pill intake over time), after having commenced supplementation with the assigned multivitamin, and the p-value was determined by the Wilcoxon (Peto-Prentice) test.

SECONDARY OUTCOMES:
The overall use of Pregvit® vs Orifer®F (adherence) | Study completion was defined as completing monthly telephone interviews (when possible) to document pill intake and adverse events up until the end of pregnancy (i.e. 36 weeks gestation or further).
  Rates of adherence and adverse events will be compared by using chi-squared tests, as appropriate. Adherence will be also compared between the 2 treatment groups through Kaplan-Meier survival curves in 2 ways. The second survival curve analysis will compare overall adherence among women who commenced supplementation with the assigned multivitamin, at any percentage of pill intake over time, and the p-value was determined by the log rank statistic. All curves will be plotted from the coordinates of 100% (y-axis point of 1.0) at time zero (x-axis point of 0) to represent that at the beginning of the study, all subjects who commenced supplementation in each multivitamin group were adherent.
The rates of overall adverse events and specific side effects between the two groups | Study completion was defined as completing monthly telephone interviews (when possible) to document pill intake and adverse events up until the end of pregnancy (i.e. 36 weeks gestation or further).
  Rates of adherence and adverse events will be compared by using chi-squared tests, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Koren, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- See also: Effect of iron content on the tolerability of prenatal multivitamins in pregnancy — http://www.ncbi.nlm.nih.gov/pubmed/18482454
- See also: Adherence and tolerability of iron-containing prenatal multivitamins in pregnant women with pre-existing gastrointestinal conditions. — http://www.ncbi.nlm.nih.gov/pubmed/19757261